CLINICAL TRIAL: NCT01233674
Title: Examination of Left Atrial Fibrosis Using MRI
Status: Withdrawn | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 08120067
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2016-01

CONDITIONS: Fibrosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- patients referred for standard of care MRI

SUMMARY:
This study evaluates images obtained from a standard clinical cardiac MRI for evidence of fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* being scheduled for a standard of care MRI

Exclusion Criteria:

- patient unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients referred for standard of care MRI
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC CVI, Pittsburgh, Pennsylvania, United States